CLINICAL TRIAL: NCT02037789
Title: A Retrospective Study to Identify New "Omics" Biomarkers of Chronic/Persistent Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: GENOS (Other); Ip Research Consulting Sasu (Industry); Helmholtz Zentrum München (Industry); YURII AULCHENKO (Unknown); King's College London (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: Pain-OMICS RT
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Persistent/Chronic Low Back Pain
Keywords: pain; low back pain; GWAS; glycomics; activomics
MeSH Terms: conditions — Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected from cases (patients already diagnosed with persistent/chronic low back pain) and from controls (healthy subjects).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Low back pain (LBP) is one of the most common medical problems encountered in daily life; it is related to disability and work absence and accounts for high economical costs in Western societies.

Low-back pain is a diverse group of mixed pain syndromes (neuropathic and nociceptive) with different molecular pathologies at different structural levels displaying similar clinical manifestations. Currently, there are limited biomarkers (mostly imaging) or clinical findings that can be used objectively to help the physician in precise anatomic diagnosis leading to the safest and most cost-effective treatment for the patient (reduction of direct and indirect costs and improvement of treatment efficacy).

The main aim of this trial is to identify all "omics biomarkers" associated with susceptibility to chronic/persistent LBP and its different pathophysiology.

DETAILED DESCRIPTION:
Retrospective observational multinational clinical study, with a case control design.

Investigators will compare "omic biomarkers" between patients with and without persistent chronic low back pain (CLBP).

"OMIC" biomarkers investigated will be genetics, glycomics and activomic. Genetics through GWA studies has already obtained important results in pain research; however concerning low back pain, there is not yet suitable genotype-phenotype correlations helpful to stratify patients.

Glycomics is an emerging field that has recently been identified as a priority for the next decade by the US National Academies of Science. Many common complex diseases will be associated with specific changes in glycan structures. In addition, common genetic polymorphisms influencing glycosylation and consequent differences in glycome composition could be important diagnostic and prognostic markers. The first studies reporting protein glycosylation in large human population samples have been recently published by partners in the consortium. Reliable identification of valid associations between specific glyco-phenotypes and predisposition for the development or progression of a specific disease requires analysis of thousands of patients.

Activomics: combines data about enzymatic activity of numerous numerous post-translational modification proteins in an integrated model which provides dynamic characterization of the current state of an organism. In this project information about numerous proteases, kinases, phosphatases and glycosidases will be collected and used to complement the existing phenotype information.

ELIGIBILITY:
Inclusion Criteria of patients with persistent CLBP:

* age: older than 18;
* chronic/persistent pain (pain lasting longer than 12 weeks) between the costal margins and gluteal fold, with or without symptoms into one or both legs
* written informed consent signed;
* Caucasian ancestry

Inclusion Criteria of healthy volunteers:

* age: older than 18;
* without any chronic/persistent pain (pain lasting longer than 12 weeks) in the last one year;
* written informed consent signed;
* Caucasian ancestry

Exclusion Criteria:

* evidence of clinically unstable disease;
* severe psychiatric disorder (excluding mild depression) or mental impairment;
* recent history ( < 1 year) of spinal fracture;
* pain in the back due to spinal tumor or infection;
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will be collected at each participating centre. Every effort will be made to accumulate a well phenotyped cohort of patients with persistent CLBP, sub-grouped into 6 categories: discogenic pain, spinal stenosis (congenital or acquired), facet joint pain, sacroiliac joint pain, low back pain with radicular pain (not predominant radicular pain) and widespread low back pain.
  Controls (patients without chronic/persistent pain as defined above) will be retrieved from 2 different sources:
  Existing biobanks of healthy subjects which have collected information about chronic/persistent back pain.
  Subjects from the companion prospective study on acute LBP who will not have developed CLBP.
  Age (decades) and gender distribution of controls will be similar to cases.
Sampling Method: Non-Probability Sample
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
GENETIC OUTCOME | 30 months
  The primary objective is to recognize genetic variants associated with persistent CLBP patients compared to patients without chronic/persistent pain. Through a Genetic Wide Association Study (GWAS) investigators will correlate genetic variants associated with persistent CLBP in a wide, international population of European ancestry.

SECONDARY OUTCOMES:
GLYCOMIC AND ACTIVOMIC OUTCOME | 30 months
  Recognize Glycomic and Activomic data associated with persistent CLBP patients compared to patients without chronic/persistent pain. The sample size will better defined after the first interim analysis of first 400 patients.
STRATIFICATION OF OUR POPULATION | 30 months
  All "omic" data will be compared stratifying our population according to:
  * Pathophysiology: discogenic pain, spinal stenosis, facet joint pain, sacroiliac joint pain, low back pain with radicular pain (not predominant radicular pain) and widespread pain.
  * pain intensity
  * response to treatment
  * duration of pain

CONTACTS AND LOCATIONS:
Overall Officials: MASSIMO ALLEGRI, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (6):
- The Center for Clinical Research (CPI), Winston-Salem, North Carolina, United States
- Edith Cowan University (ECU), Perth, Australia
- Multidisciplinary Pain Centre, Hospital Oost-Limburg (ZOL), Genk, Belgium
- "St.Catharine" Orthopedics, Surgery, Neurology and Physical Medicine and Rehabilitation Specialty Hospital (St-Cat), Zabok, Croatia
- Italy (2):
  - Anesthesia and Pain Therapy Department, Università degli Studi di Parma (UNIPR), Parma
  - Fondazione IRCCS Policlinico San Matteo (OSM), Pavia

REFERENCES:
- [Derived] Allegri M, De Gregori M, Minella CE, Klersy C, Wang W, Sim M, Gieger C, Manz J, Pemberton IK, MacDougall J, Williams FM, Van Zundert J, Buyse K, Lauc G, Gudelj I, Primorac D, Skelin A, Aulchenko YS, Karssen LC, Kapural L, Rauck R, Fanelli G; PainOMICS Group. 'Omics' biomarkers associated with chronic low back pain: protocol of a retrospective longitudinal study. BMJ Open. 2016 Oct 19;6(10):e012070. doi: 10.1136/bmjopen-2016-012070. PMID 27798002